CLINICAL TRIAL: NCT06928428
Title: Metacognitive Therapy for Depression and Generalized Anxiety Disorder in Primary Health Care, Feasibility of a Blended Mediated Treatment
Brief Title: Metacognitive Therapy for Depression and Generalized Anxiety Disorder in Primary Care, Blended Version of Mediated Treatment
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Region Stockholm (Other Government)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: FoUI-990130
Record Dates: First submitted 2024-10-02; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-03

CONDITIONS: Depression NOS; Generalized Anxiety Disorder
Keywords: primary care; depression; generalized anxiety disorder; metacognitive therapy; blended treatment
MeSH Terms: conditions — Depression; Generalized Anxiety Disorder

STUDY DESIGN:
Intervention Model Description: Study 1: Feasibility will be performed in single group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Blended metacognitive therapy (bMCT) (Experimental): Blended metacognitive therapy (bMCT): New about this treatment is that it is given both via the internet and through meetings with a therapist. Participants work with the treatment independently via an internet platform and meet their therapist for therapy sessions up to 6 times during the course of the treatment.
  Interventions: Behavioral: Metacognitive therapy, blended format

INTERVENTIONS:
Behavioral: Metacognitive therapy, blended format — Blended metacognitive therapy (bMCT): New about this treatment is that it is given both via the internet and through meetings with a therapist. Participants work with the treatment independently via an internet platform and meets their therapist for therapy sessions up to 6 times during the course of the treatment. Key components of the original manual are retained, but adapted to better fit the digital format. A handbook for therapists is developed to facilitate the implementation of the blended format and optimize execution. The digital parts of the treatment for depression and GAD consist of 10 interactive modules located in the Support and Treatment (SoB) platform. The sessions are divided in a flexible way between physical and digital sessions that therapist and patient agree on. The patient has access to all modules but receive instructions from their therapist which module is relevant for each week. During the treatment, the patient can write text messages to his/her therapist.

SUMMARY:
The goal of this clinical trial is to investigate a new format of metacognitive therapy (MCT) for primary care patients with depression or generalized anxiety disorder (GAD) called blended MCT (bMCT). What is new about bMCT is that it is given both via the internet and through meetings with a therapist. In this study, we first want to investigate if it is feasible to deliver bMCT in primary health care to patients with depression or GAD. Secondly, we want to investigate whether the format of bMCT can provide as good treatment effects as only personally mediated MCT.

The content of both formats of treatment is based on MCT methods for depression and GAD which have shown to be effective in previous research studies. bMCT means to work with the treatment independently via an internet platform and to meet the therapist for therapy sessions up to 6 times during the course of the treatment. Meetings will take place at the primary care center or via video call. As part of the treatment are mediated via the internet, participants need to have access to an Internet-connected computer/electronic device and be able to work with the material about 3 hours per week during the course of the treatment. Standard MCT involves seeing the therapist for 8-12 treatment sessions at the primary care center or via video call.

In the first study, all patients diagnosed with depression or GAD at Liljeholmen primary care center, after giving informed consent, will receive bMCT. In the second study, more primary health care centers will be involved and participants will be randomly allocated to either bMCT or standard MCT.

The active treatment lasts for 8-12 weeks. The treatment is estimated to involve approximately 3 hours of therapy work per week. Participants will be asked to fill in questionnaires before the treatment, weekly during the treatment, immediately after the treatment (post-treatment) and follow-ups at 6 and 12 months after post-treatment. The forms contain questions about your well-being, background and experience of the treatment. Filling in questionnaires is estimated to take 30 minutes on four measurement occasions. Participating also means giving permission for treatment conversations to be audio recorded. The recording is coded so that independent assessors can examine the therapists' competence, and see that the therapists follow the instructions for the current treatment method.

DETAILED DESCRIPTION:
Study 1. Feasibility study: Outcome measures of acceptability, feasibility and compliance:

a. What percentage of surveyed patients choose to participate in bMCT? b. What is the dropout rate, given reasons for dropping out? c. How many modules do the patients complete, from 1 to 8? d. patient satisfaction with treatment (Client Satisfaction Questionnaire, CSQ-8, range from 8 low satisfaction to 32 high satisfaction) d. Any reported negative effects of treatment e. Adherence and competence in delivering MCT sessions (MCT-Competence Scale, MCT-CS, 18 items, scale 0-5)

Study1: Experience and Usability, qualitative method:

1. How are bMCT and treatment materials experienced by patients and therapists respectively?
2. What facilitates and hinders the implementation of bMCT?

Study1: Preliminary clinical effects:

1. symptoms of depression (PHQ-9, 0-27), symptoms of GAD (PSWQ, 16-80)
2. quality of life (5-item Satisfaction with Life Scale, SWLS, 0-35)

d. functional level (WHO Disability Assessment Schedule 2.0, WHODAS, 0-48) e. self-assessed ability to work (Work Ability Index, WAI 0-10)

Study 2: randomized controlled study, additional measurements of acceptability, feasibility, compliance: Varies

1. proportion completed modules between groups?
2. percentage dropouts between groups?
3. therapist competence and adherence to MCT between groups?
4. patient satisfaction with treatment (CSQ-8, range from 8 low satisfaction to 32 high satisfaction)

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed depressive episode/recurrent depression (ICD code F32., F33.), or generalized anxiety disorder (ICD code F41.1) as primary diagnosis
* Informed consent
* Access to the internet
* Age ≥18 years
* In the event of psychopharmaceutical medication (e.g. antidepressants), the dosage must have been stable at least 4 years before inclusion

Exclusion Criteria:

* Other psychiatric condition in need of immediate treatment and/or assessed to be the patient's primary problem (e.g. bipolar disorder, psychosis, alcohol or substance use syndrome or severe eating disorder),
* Other ongoing psychological treatment
* Insufficient knowledge of the Swedish language (e.g. that an interpreter is needed during patient visits), cognitive failure or insufficient computer skills to be able to assimilate the text-based digital part of the treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Acceptability, is bMCT an acceptable treatment for primary care patients with depression or GAD? | Measurements are delivered at enrollment before treatment, during treatment week 1 to 12, and post-treatment after 12 weeks.
  What percentage of surveyed patients choose to participate in bMCT? Measured as percentage of surveyed and eligible patients with a diagnosis of depression or GAD who agree to participate in the treatment study.
Adherence, do the participating patients fulfill the bMCT modules? | Measurements are delivered at enrollment pre-treatment, post-treatment when treatment is finished after 10 weeks (treatment range 6 to maximum of 12 treatment sessions), six months after post-treatment, and 12 months after post-treatment.
  How many modules in the bMCT protocol do the patients complete, from 1 to 8? Measured by number of gathered patient-reported assignments, one for each module out of eight in the SoB-portal.
What is the dropout rate of included patients in bMCT? | Measurements are reported during treatment if interrupted and summarized post-treatment when treatment is finished after 10 weeks (treatment range 6 to maximum of 12 treatment sessions).
  Dropout rate is measured as percentage of included patients who choose to drop out before the completion of bMCT treatment.
Satisfaction with bMCT treatment | Measurements are delivered at post-treatment when treatment is finished after 10 weeks (treatment range 6 to maximum of 12 treatment sessions).
  Patient satisfaction with treatment will be measured with the Client Satisfaction Questionnaire, CSQ-8, which ranges from 8 "low satisfaction" to 32 "high satisfaction" with treatment.
Any reported negative effects of bMCT? | Measurements are delivered at post-treatment when treatment is finished after 10 weeks (treatment range 6 to maximum of 12 treatment sessions).
  Measured with the Negative Effects Questionnaire, NEQ, 32 items where participating patients report on a Likert scale 0 to 4, thus, a total range of 0 "no reported negative effects" to 128 "maximum reported negative effects".
The therapists' competence in carrying out the bMCT treatment | Sessions are audio-recorded during treatment week 1 to 12, assessments of the recordings are carried out post-treatment after 12 weeks up to 6 months post-treatment.
  All treatment sessions are audio-recorded. For each therapist three randomly selected recordings are assessed for a total score on the Metacognitive Therapy Competence Scale, MCT-CS, witch includes 18 items and rates competence on a Likert scale that ranges from 0 "not done, not applicable " to 5 "very good level", thus, a total scale ranging from 0 to 90. Assessments are performed by external independent expert assessors with deep knowledge of MCT and prior experience in using the MCT-CS scale.
Patients experience of bMCT, qualitative method | Interviews are carried out post-treatment when treatment is finished after 10 weeks up to two months post treatment (treatment range 6 to maximum of 12 treatment sessions).
  Individual semi structured interviews are performed with a selection of participating patients post treatment with questions about their experiences of bMCT. Interviews are audio-recorded and transcribed verbatim for qualitative content analysis.
Therapists' experience of carrying out bMCT, qualitative method | Focus group discussion with participating therapists is carried out post treatment when all patients in the feasibility study have finished treatment 12 weeks up to 6 months post treatment.
  Focus group interview with participating therapists. Semi structured questions and discussions about their experiences of mediating bMCT. Audio-recorded discussions are transcribed and analyzed with qualitative content analysis.
What facilitates the implementation of bMCT? Qualitative method | Interviews with patients are carried out post-treatment after 12 weeks up to two months post treatment. Focus group with therapists when all patients in the feasibility study have finished treatment 12 weeks up to 6 months post treatment.
  Individual interviews with a selection of participating patients and focus group interview with participating therapists. Semi structured questions about perceived facilitators of bMCT. Audio-recorded discussions are transcribed and analyzed with qualitative content analysis.
What hinders the implementation of bMCT? Qualitative method | Interviews with patients are carried out post-treatment, after 12 weeks, and focus group with therapists when all patients in the feasibility study have finished treatment 12 weeks up to 6 months post treatment.
  Individual interviews with a selection of participating patients and focus group interview with participating therapists. Semi structured questions about perceived hindering factors of bMCT. Audio-recorded discussions are transcribed and analyzed with qualitative content analysis.

SECONDARY OUTCOMES:
Preliminary clinical effects of bMCT, change in depressive symptoms | Measurements are delivered at enrollment pre-treatment, post-treatment when treatment is finished after 10 weeks (treatment range 6 to maximum of 12 treatment sessions), six months efter post-treatment, and 12 months after post-treatment.
  Preliminary clinical effects of bMCT regarding change in depressive symptoms measured with Patient Health Questionnaire-9 items, PHQ-9, range from 0 "no depressive symptoms" to 27 "severe depressive symptoms"
Preliminary clinical effects of bMCT, change in symptoms of generalized anxiety disorder (GAD) | Measurements are delivered at enrollment pre-treatment, post-treatment when treatment is finished after 10 weeks (treatment range 6 to maximum of 12 treatment sessions), six months efter post-treatment, and 12 months after post-treatment.
  Preliminary clinical effects of bMCT regarding change in symptoms of GAD measured with Penn State Worry Questionnaire, PSWQ, with a total range from 16 "no GAD symptoms" to 80 "severe GAD symptoms"
Preliminary clinical effects of bMCT, change in quality of life | Measurements are delivered at enrollment pre-treatment, post-treatment when treatment is finished after 10 weeks (treatment range 6 to maximum of 12 treatment sessions), six months efter post-treatment, and 12 months after post-treatment.
  Preliminary clinical effects of bMCT regarding change in patient rated quality of life, measured with the 5-item Satisfaction with Life Scale, SWLS. The total score ranges from 5 "extremely dissatisfied" to 35 "extremely satisfied".
Preliminary clinical effects of bMCT, change in functional level | Measurements are delivered at enrollment pre-treatment, post-treatment when treatment is finished after 10 weeks (treatment range 6 to maximum of 12 treatment sessions), six months efter post-treatment, and 12 months after post-treatment.
  Preliminary clinical effects of bMCT regarding change in patient rated functional level measured with WHO Disability Assessment Schedule 2.0, with 12 items and a total range from 0 "no impairment" to 48 "severe impairment in all daily activities".
Preliminary clinical effects of bMCT, self-assessed ability to work | Measurements are delivered at enrollment pre-treatment, post-treatment when treatment is finished after 10 weeks (treatment range 6 to maximum of 12 treatment sessions), six months efter post-treatment, and 12 months after post-treatment.
  Preliminary clinical effects of bMCT regarding change in self-assessed ability to work measured with Work Ability Index, WAI, a total range from 0 "no ability to work" to 10 "my work ability is at it's best"
Preliminary clinical effects of bMCT, change in symptoms of insomnia | Measurements are delivered at enrollment pre-treatment, post-treatment when treatment is finished after 10 weeks (treatment range 6 to maximum of 12 treatment sessions), six months efter post-treatment, and 12 months after post-treatment.
  Preliminary clinical effects of bMCT regarding change in symptoms of insomnia measured with Insomnia Severity Index, ISI, 5 items with a total range of 0 "no signs of insomnia" to 28 "severe clinical insomnia"

CONTACTS AND LOCATIONS:
Overall Officials: Sandra af Winklerfelt Hammarberg, MD, PhD, Principal Investigator — Region Stockholm and Karolinska Institutet
Locations (1):
- Liljeholmen primary care center, Academic Primary care center, SLSO, Region Stockholm, Stockholm, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: No
Due to legal reasons in Sweden we are not able to share IPD, but we will try to give access for other researchers to anonymized data upon legitimate request.

REFERENCES:
- [Background] Eldridge SM, Lancaster GA, Campbell MJ, Thabane L, Hopewell S, Coleman CL, Bond CM. Defining Feasibility and Pilot Studies in Preparation for Randomised Controlled Trials: Development of a Conceptual Framework. PLoS One. 2016 Mar 15;11(3):e0150205. doi: 10.1371/journal.pone.0150205. eCollection 2016. PMID 26978655
- [Background] Cuijpers P, Berking M, Andersson G, Quigley L, Kleiboer A, Dobson KS. A meta-analysis of cognitive-behavioural therapy for adult depression, alone and in comparison with other treatments. Can J Psychiatry. 2013 Jul;58(7):376-85. doi: 10.1177/070674371305800702. PMID 23870719
- [Background] van der Heiden C, Muris P, van der Molen HT. Randomized controlled trial on the effectiveness of metacognitive therapy and intolerance-of-uncertainty therapy for generalized anxiety disorder. Behav Res Ther. 2012 Feb;50(2):100-9. doi: 10.1016/j.brat.2011.12.005. Epub 2011 Dec 21. PMID 22222208
- [Background] Andersson G, Titov N, Dear BF, Rozental A, Carlbring P. Internet-delivered psychological treatments: from innovation to implementation. World Psychiatry. 2019 Feb;18(1):20-28. doi: 10.1002/wps.20610. PMID 30600624
- [Background] Hedman E, Ljotsson B, Lindefors N. Cognitive behavior therapy via the Internet: a systematic review of applications, clinical efficacy and cost-effectiveness. Expert Rev Pharmacoecon Outcomes Res. 2012 Dec;12(6):745-64. doi: 10.1586/erp.12.67. PMID 23252357
- [Background] Af Winklerfelt Hammarberg S, Toth-Pal E, Jansson-Frojmark M, Lundgren T, Westman J, Bohman B. Intolerance-of-uncertainty therapy versus metacognitive therapy for generalized anxiety disorder in primary health care: A randomized controlled pilot trial. PLoS One. 2023 Jun 14;18(6):e0287171. doi: 10.1371/journal.pone.0287171. eCollection 2023. PMID 37315099
- [Background] Cuijpers P, Donker T, van Straten A, Li J, Andersson G. Is guided self-help as effective as face-to-face psychotherapy for depression and anxiety disorders? A systematic review and meta-analysis of comparative outcome studies. Psychol Med. 2010 Dec;40(12):1943-57. doi: 10.1017/S0033291710000772. Epub 2010 Apr 21. PMID 20406528